CLINICAL TRIAL: NCT02057588
Title: Enhanced Diagnosis of Ventricular Activation Pattern Using Intracardiac Electrograms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR-12-082-FR-HV
Record Dates: First submitted 2014-01-31; First posted 2014-02-07 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Arrythmia
Keywords: ablation
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LV Paced sites (Other): LV pacing sites : Patients will be paced from various left ventricular origin, defined by their 3D localization.
  Interventions: Procedure: LV pacing site

INTERVENTIONS:
Procedure: LV pacing site — Patient will be paced in VVI mode from Left ventricle specific position for a short period of time per position in order to cover spontaneous ventricular activity

SUMMARY:
The objective of this study will be to evaluate the ability of IEGMs (Signal recorded from implanted pacing leads) and pseudo ECGs (derived from various IEGMs) to characterize various electrical conduction patterns. Electroanatomic mapping data and 12 Lead ECG will also be collected to characterize electrical conduction patterns during standard electrophysiology exam.

ELIGIBILITY:
Inclusion Criteria:

* Patient with SJM CRM device implanted for more than 90 days

Exclusion Criteria:

* Suspicion of lead dislodgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Correlation of ventricular activation patterns determined by 12-lead ECG and device IEGMs-based method | Acute, intraoperative
  Correlation coefficient between ventricular activation patterns determined by a traditional technique, 12-lead ECG based vs. device based IEGMs method.

SECONDARY OUTCOMES:
Ventricular activation origin location determined by IEGMs based method vs. by detailed mapping | Acute, intraoperative
  Use of available IEGMs recorded on implanted device to discriminate specific VT origin and pattern and compare the results to the detailed mapping data

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Sacher, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU haut leveque, Pessac, France